CLINICAL TRIAL: NCT06763159
Title: A Phase I, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of HS-20124 in Patients with Advanced Solid Tumors
Brief Title: A Study of HS-20124 in Patients with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20124-101
Record Dates: First submitted 2024-11-08; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Solid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HS-20124 (Phase Ia：Dose escalation ) (Experimental): HS-20124 for IV infusion of various dose strengths administered in 21 day dosing cycles
  Interventions: Drug: HS-20124 (Phase Ia：Dose escalation )
- HS-20124 (Phase Ib: Dose expansion) (Experimental): The recommended dose from the dose-escalation stage and other potential doses will be further explored
  Interventions: Drug: HS-20124 (Phase Ib: Dose expansion)

INTERVENTIONS:
Drug: HS-20124 (Phase Ia：Dose escalation ) — Participants will receive HS-20124 in 21 day dosing cycles. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Arms: HS-20124 (Phase Ia：Dose escalation )
Drug: HS-20124 (Phase Ib: Dose expansion) — Participants will receive HS-20124 in 21 day dosing cycles. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Arms: HS-20124 (Phase Ib: Dose expansion)

SUMMARY:
HS-20124 is a novel DAR-8 antibody-drug conjugate （ADC） targeting CDH6. In preclinical studies, it inhibited tumor cell growth expressing CDH6 in vitro and in vivo. The first-in-human trial is conducted to assess the maximum tolerated dose (MTD) and dose limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of HS-20124 in Patients With Advanced Solid Tumors.

DETAILED DESCRIPTION:
This is a Phase 1a/1b open-label, multicenter study with dose escalation and dose expansion cohorts to evaluate the safety, tolerability, PK and preliminary efficacy of HS-20124 in patients with advanced solid tumors.

The dose escalation will utilize rolling-6 design. In phase of dose expansion, preliminary efficacy will be evaluated in planned expansion cohorts that include patients with specific advanced solid tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. At least age of 18 years at screening;
2. Histologically or cytologically confirmed, locally advanced or metastatic solid tumors for which standard treatment either does not exist or has proven ineffective or unavailable or intolerable
3. At least one extra-cranial measurable lesion according to RECIST 1
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1
5. Life expectancy >= 12 weeks
6. Men or women should be using adequate contraceptive measures throughout the study;
7. Females subjects must not be pregnant at screening or have evidence of non-childbearing potential
8. Signed and dated Informed Consent Form

Exclusion Criteria:

1.Treatment with any of the following:

1. Previous or current treatment with CDH6 targeted therapy
2. Any cytotoxic chemotherapy and small molecule targeted anticancer drugs within 21 days or five half-livesprior to the first scheduled dose of HS-20124
3. Prior treatment with a monoclonal antibody or investigational agents within 28 days prior to the first scheduled dose of HS-20124
4. Radiotherapy with a limited field of radiation for palliation within 2 weeks, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks prior to the first scheduled dose of HS-20124
5. Major surgery within 4 weeks prior to the first scheduled dose of HS-20124 2. Subjects with previous or concurrent malignancies 3. Inadequate bone marrow reserve or organ dysfunction 4. Evidence of cardiovascular risk 5. Evidence of current severe or uncontrolled systemic diseases 6. Evidence of mucosal or internal bleeding within 1 month prior to the first scheduled dose of HS-20124 7. Severe infection within 4 weeks prior to the first scheduled dose of HS-20124 8. Subjects with current infectious diseases 9. History of neuropathy or mental disorders 10. Pregnant or lactating female 11. History of severe hypersensitivity reaction, severe infusion reaction or idiosyncrasy to drugs chemically related to HS-20124 or any of the components of HS-20124

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of complete response (CR) an | 3 weeks after initiation of treatment
  To determine the MTD/MAD for further evaluation of IV administration of HS-20124 in subjects with advanced solid tumors
Ⅰb (Dose-Expansion Stage): Objective response rate (ORR) determined by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | From the first dose up to PD or withdrawal from study, whichever came first.
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of complete response (CR) and partial response (PR) [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)]

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | From the first dose through 30 days post end of treatment
  AE assessed by investigator exclusively related to subject's underlying disease or medical condition [graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0]. Any untoward medical occurrence in a clinical study participant, whether or not considered related to the medicinal product. Incidence and severity of AEs are assessed according to vital signs, laboratory variables, physical examination, electrocardiogram, etc.
Observed maximum plasma concentration (Cmax) | At the end of Cycle 1 (each cycle is 21 days)
  Cmax will be obtained following administration of the first dose of HS-20124 during the first cycle
Time to reach maximum plasma concentration (Tmax) | At the end of Cycle 1 (each cycle is 21 days)
  Tmax will be obtained following administration of the first dose of HS-20124 during the first cycle
Terminal half-life (T1/2) | At the end of Cycle 1 (each cycle is 21 days)
  Apparent terminal half-life is the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by λz.
Percentage of participants with antibodies to HS-20124 in serum | At the end of Cycle 1 (each cycle is 21 days)
  Serum samples were collected for the determination of anti-drug antibody (ADA) at designated time points
ORR determined by investigators according to RECIST 1.1 (dose-escalation stage) | during the intervention
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of CR and PR (Confirmed CR/PR assessment require at least 1 repeat).
Duration of response (DOR) determined by investigators according to RECIST 1.1 | during the intervention
  DoR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].
Progression-free survival (PFS) determined by investigators according to RECIST 1.1 | From the randomization/first dose up to PD or death, whichever came first
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). PFS was defined as the time from random assignment (dose expansion stage) or first dose (dose escalation stage) to PD or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality, China